CLINICAL TRIAL: NCT06405451
Title: Pilot Experimental Study on the Impact of a Respiratory Muscle Training Program in Patients With Multiple Sclerosis
Brief Title: Respiratory Muscle Training Program in Patients With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Collaborators: Fundación Madrid contra la Esclerosis Múltiple (FEMM) (Unknown); Sanitas (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 23/685-E
Record Dates: First submitted 2024-04-08; First posted 2024-05-08 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2024-02

CONDITIONS: Multiple Sclerosis; Respiration Disorders
Keywords: multiple sclerosis; treatment; trunk disorder; balance; respiratory function
MeSH Terms: conditions — Multiple Sclerosis; Respiration Disorders; Respiratory Aspiration

STUDY DESIGN:
Intervention Model Description: This is a quasi-experimental pre-post trial. The research will be conducted in accordance with the Helsinki Declaration and the Personal Data Protection and Guarantee of Digital Rights Act (Organic Law 3/2018). The design of this project will adhere to the standard protocol elements of a clinical trial: SPIRIT statement.
Who Masked: Outcomes Assessor
Masking Description: Blinding will involve the evaluators, who will be unaware of which intervention group each subject belongs to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment (Active Comparator): Conventional treatment to improve trunk control and stability for 30 minutes, twice a day, six times a week.
  Interventions: Other: Conventional treatment
- Experimental treatment (Experimental): Respiratory muscle training will be conducted using the Threshold IMT-Philips inspiratory training device and the Threshold PEP expiratory training device, both from Respironics®. Participants will be comfortably seated in a chair with their feet on the ground, without back support, and with the trunk at a 90° angle to the hips. A conventional nasal clip will be used to prevent air leaks. During forced expiratory training, participants will use the ThresholdPEP® with a customized mouthpiece and perform forced expiration through the resistance device. Inspiratory muscle training will follow the same procedure using the Threshold IMT®. Both inspiratory and expiratory training will be repeated 10-15 times, 5 sets for 20 minutes in one session, with a rest time of 30-60 seconds between each set.
  Interventions: Other: Conventional treatment; Other: Experimental treatment

INTERVENTIONS:
Other: Conventional treatment — Conventional treatment to improve trunk control and stability for 30 minutes, twice a day, and six times per week.
Other: Experimental treatment — Respiratory muscle training will be conducted using the Threshold IMT-Philips inspiratory training device and the Threshold PEP expiratory training device, both from Respironics®. Participants will be comfortably seated in a chair with their feet on the ground, without back support, and with the trunk at a 90° angle to the hips. A conventional nasal clip will be used to prevent air leaks. During forced expiratory training, participants will use the ThresholdPEP® with a customized mouthpiece and perform forced expiration through the resistance device. Inspiratory muscle training will follow the same procedure using the Threshold IMT® (45).
  Both inspiratory and expiratory trainings will be repeated 10-15 times, 5 sets for 20 minutes in one session, with a rest time of 30-60 seconds between each set.
  Arms: Experimental treatment

SUMMARY:
This is a quasi-experimental pre-post trial aimed at investigating the effects of respiratory muscle training (RMT) as trunk stabilization exercise in patients diagnosed with multiple sclerosis (MS)

DETAILED DESCRIPTION:
Multiple sclerosis (MS) is a chronic disease of the central nervous system that can affect various bodily functions, including the respiratory muscles. Weakness in these muscles can lead to a range of complications, including impacting trunk stability, which may result in difficulties maintaining a balanced and stable posture.

While the impact of MS on respiratory muscles and trunk stability is an area of interest in medical research, a definitive consensus on the efficacy of respiratory muscle training (RMT) to improve trunk stability in MS patients has not yet been reached. Several studies have yielded mixed results, leading to uncertainty regarding the effectiveness of this specific intervention.

The complex nature of multiple sclerosis necessitates a multidisciplinary approach to address its various clinical manifestations. In addition to pharmacological treatment, physical and occupational therapy play a crucial role in symptom management and improving patients' quality of life. Although respiratory muscle training may offer potential benefits, further research and well-designed clinical trials are needed to determine its effectiveness and role in the comprehensive management of trunk stability in MS patients.

- General objective: The aim of this study is to investigate the effects of respiratory muscle training (RMT) as a trunk stabilization exercise in patients diagnosed with multiple sclerosis (MS).

- Specific objectives: To analyze the effects of RMT on lung function measured through spirometric tests.

To evaluate the effect of RMT on respiratory muscle strength using maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP).

To investigate the changes produced by RMT on abdominal and diaphragmatic muscle structures measured through ultrasound.

To analyze the effect of RMT on trunk control measured with the Trunk Impairment Scale (TIS).

To study the effect of RMT on balance assessed with the Berg Balance Scale (BBS).

To investigate the effect of RMT on gait capacity and transfers evaluated through the Timed Up and Go (TUG) test.

- Study design: This is a quasi-experimental pre-post trial. The research will be conducted following the principles outlined in the Helsinki Declaration and the Personal Data Protection and Guarantee of Digital Rights Act. The conception of this project will follow the standard elements defined in the SPIRIT (Standard Protocol Items: Recommendations for Interventional Trials) statement.

- Sample size: Sample size calculation will be based on data obtained from a pilot study involving 20 subjects. Subsequently, G*POWER software will be used to calculate the sample size using data obtained for the main variable expressed through diaphragm thickness to determine the effect size. Throughout the project, a power of 80%, an alpha error of 0.05 (one-tailed), and a 95% confidence interval will be employed.

- Subjects: Subjects will be recruited through a previously signed agreement with the Multiple Sclerosis Patients Association, the European University of Madrid, and Sanitas. Subjects will belong to the Multiple Sclerosis Patients Association, and sessions will be conducted at Sanitas centers in Madrid affiliated with the agreement.

- Inclusion criteria: Age between 18 and 70 years. Confirmed diagnosis of Multiple Sclerosis based on McDonald's criteria, with a disease duration of more than two years (relapsing or progressive).

All multiple sclerosis patients according to the Expanded Disability Status Scale (EDSS) will be included.

Stable medical treatment for at least six months prior to the intervention. Absence of cognitive impairment, with the ability to understand instructions and achieve a score equal to or greater than 24 on the Mini-Mental State Examination.

*All wheelchair-bound and non-wheelchair-bound patients will be included, as both groups may benefit from the intervention due to increased trunk motor control. However, only subjects capable of walking will undergo walking-related variables or tests (up to 6 on the EDSS scale).

- Exclusion criteria: Diagnosis of another neurological disease or musculoskeletal disorder other than MS.

Diagnosis of any cardiovascular, respiratory, or metabolic disease, or other conditions that may interfere with this study.

Exacerbation or hospitalization in the last three months before initiating the assessment protocol, or during the therapeutic intervention process.

Receiving a cycle of steroids, intravenously or orally, six months before the start of the assessment protocol and within the intervention period of the study duration.

- Variables, measurements, and measurement instruments: Pulmonary function: forced vital capacity (FVC), forced expiratory volume in one second (FEV1) will be obtained.

Muscle strength, MIP and MEP variables: maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP) will be measured.

Ultrasound measurements: of the diaphragm (ultrasound measurement of diaphragm thickness; ultrasound measurement of diaphragm excursion), of the abdominal musculature (ultrasound measurement of abdominal diastasis and abdominal wall).

Trunk Impairment Scale (TIS): static and dynamic trunk stability will be measured.

Berg Balance Scale (BBS): patient balance will be measured. Timed Up and Go (TUG): activity limitations will be assessed. Therapeutic adherence.

- Therapetic intervention program: Before starting the therapeutic intervention protocol, patients will be informed about the study through an informed consent form (APPENDIX I), which they will sign and submit. The necessary material for conducting the intervention will also be provided, which will be delivered to the patient's home.

The therapeutic intervention program will be carried out for 30 minutes, twice a day, and six times a week, following the protocol by Lee et al.

Note: During respiratory work, patients may experience dizziness, headaches, changes in heart rate, or desaturations. Therefore, to maintain safety margins, participants will be continuously monitored with an FDA-approved fingertip pulse oximeter.

To determine the percentage of work of MIP and MEP, this variable will be taken using a Micro RPM® respiratory pressure device from Micro Medical, Kent, United Kingdom. Participants will work at 40%-60% of the maximum MIP and MEP, according to the clinical trial by Brita Klefbeck et al.

Respiratory muscle training will be performed with the Threshold IMT-Philips inspiratory training device and the Threshold PEP expiratory training device, both from Respironics®. Participants will be comfortably seated in a chair with their feet on the ground, without back support, and with the trunk at a 90° angle to the hips. A conventional nasal clip will be used to prevent air leaks. In forced expiratory training, participants will use the ThresholdPEP® with a custom mouthpiece and perform forced expiration through the resistance device. Inspiratory muscle training will follow the same procedure using the Threshold IMT®.

Both inspiratory and expiratory training will be repeated 10-15 times, 5 sets for 20 minutes in one session, with a rest time of 30-60 seconds between each set.

Patients will receive a phone call every Monday during the 6 weeks of the intervention to check if they are performing the exercises and to answer any questions arising from the training.

- Statistical methods: Qualitative variables will be expressed as absolute number and percentage, and quantitative variables as mean ± standard deviation if they follow a normal distribution, or as median and interquartile range (IQR) if not. Kolmogorov-Smirnov or Shapiro-Wilk tests (if the sample is less than 50) will be used to check the normality of data distributions.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of Multiple Sclerosis based on McDonald criteria, with a disease duration of more than two years (relapsing or progressive) (McDonald et al., 2001).
* All multiple sclerosis patients are included according to the Kurtzke Disability Status Scale (EDSS) ANEX II (Kurtzke 1983, Tollár 2020).*
* Stable medical treatment for at least the six months prior to the intervention (Tollár, 2020).
* Absence of cognitive impairment, with the ability to understand instructions and achieve a score equal to or greater than 24 on the Mini-Mental State Examination (Folstein, Folstein & McHugh, 1975, Tollár 2020).

Exclusion Criteria:

* Diagnosis of another neurological disease or musculoskeletal alteration other than MS.
* Diagnosis of any cardiovascular, respiratory, or metabolic disease, or other conditions that may interfere with this study.
* Experienced exacerbation or hospitalization within the last 3 months prior to initiating the assessment protocol, nor during the therapeutic intervention process.
* Received a cycle of steroids, intravenously or orally, 6 months prior to the start of the assessment protocol and within the study intervention period.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2024-04-09 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pulmonary function | 2 months
  Spirometric functional testing will be conducted according to SEPAR Regulation (2013). Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 second (FEV1) will be measured using a pneumotachograph or open system spirometer. Participants' birth date and height will be recorded to compare with population averages. They will sit upright in a chair, wearing loose clothing, with a nasal clip to prevent leaks. Instructions will be given to exhale fully, then inhale deeply, hold briefly, and exhale forcefully. The researcher will correct any errors. Acceptable maneuvers must start quickly, have steady exhalation, and last at least 6 seconds. Three to eight maneuvers will be performed, and the best FVC and FEV1 values will be recorded.
Respiratory muscle strength | 2 months
  Respiratory muscle strength is assessed using maximum inspiratory pressure (MIP) and maximum expiratory pressure (MEP).
  After measuring FVC and FEV1, participants will rest for 5 minutes before the next maneuver. MEP will be performed first, followed by MIP. Each maneuver will be repeated 6 times with 1 minute of rest in between. The highest MIP and MEP values, measured in cm3 of H2O, will be compared with population norms.
Abdominal and diaphragmatic muscle structure | 2 months
  Ultrasound measurements of the abdominal wall and diaphragm will be conducted by an expert using the LOGIQ S7 Expert ultrasound system. To ensure accuracy and compliance with RUSI regulations, three measurements will be taken for each parameter, then averaged.
  1. Diaphragm Ultrasound: Thickness and excursion during inspiration will be evaluated. Measurements will be taken in the right hemidiaphragm using a 10-12MHz linear probe, perpendicular to the intercostal space. Diaphragm thickness below 2mm is considered atrophy. Diaphragm excursion will be measured using a 2.5 to 3.5 MHz convex probe during tidal and forced inspirations.
  2. Abdominal Musculature Ultrasound: Muscle layers and abdominal diastasis will be assessed. Abdominal diastasis will be measured with the participant lying supine, knees bent at 90º, and arms along the body. Muscle thickness will be measured at the navel level. Measurements will be taken at quiet and forced expiration.
Trunk control | 2 months
  Measured with the TIS Scale. The aim of this scale is to measure the static and dynamic stability of the trunk in sitting position without back support. It consists of 17 items and is scored according to the validated rubric. A higher score indicates better balance, with the highest possible score being 23 points. This scale is validated for patients with multiple sclerosis.
  This scale will only be administered to those MS patients who are able to walk.
Balance | 2 months
  It will be measured with the BERG scale. This test is used to assess balance through functional abilities in standing position. It consists of 14 items to be rated from 0 to 4 (higher scores indicate better balance), with a total score of 56.
  This scale will only be administered to those MS patients who are able to walk.
Gait and transfer capacity | 2 months
  It will be measured with the Timed Up and Go test (TUG). The objective of this test is to assess activity limitations proposed by the ICF by examining the patient's ability to walk and perform transfers. The test involves rising from a chair, walking ten meters along an indoor flat corridor, turning 180º, and returning to sit back in the same chair, using the usual assistive device. The result of the test will be the total time taken from the command until the second sitting.
  This scale will only be administered to those MS patients who are able to walk.

SECONDARY OUTCOMES:
Therapeutic adherence | 2 months
  Those who complete the protocol will be part of the "completed protocol" group, and those who do not complete the entire protocol will be part of the "intention-to-treat" variable.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Europea de Madrid, Villaviciosa de Odón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No
The study data will remain in a repository and will be available upon request from the plaintiffs.